CLINICAL TRIAL: NCT04344782
Title: Cohort Multiple Randomized Controlled Trials Open-label of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients CORIMUNO-19- BEVA Trial
Brief Title: Trial Evaluating Efficacy and Safety of Bevacizumab (Avastin®/Zeribev®) in Patients With COVID-19 Infection, Nested in the Corimmuno-19 Cohort
Acronym: CORIMMUNO-BEVA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200389-7
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: COVID19 Pneumonia
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab Injection
- Standard of Care (No Intervention)

INTERVENTIONS:
Drug: Bevacizumab Injection — Treatment includes the administration on day 1 (D1) of an infusion of Bevacizumab 7.5 mg / kg in 100 ml saline for all patients weighing 100 kg or more. In control arm, patient receives standard care.
  Arms: Bevacizumab

SUMMARY:
Bevacizumab, ZERIBEV® (Pfizer)/AVASTIN® (Roche) 25 mg/ml ®, is a recombinant humanised monoclonal IgG1 antibody It seems interesting to use bevacizumab in severe patients infected with SARS-CoV-2 requiring hospitalization in conventional unit or in ICU.

This protocol CORIMUNO19-BEVA will evaluate the efficacy and safety of AVASTIN®/ ZERIBEV® (bevacizumab) COVID-19 patients hospitalized in conventional units.

This phase 2 randomized clinical trial aimed at evaluating the efficacy and safety of AVASTIN®/ ZERIBEV® (bevacizumab) alone versus standard of care (SoC) in patients hospitalized in conventional units.

ELIGIBILITY:
Inclusion Criteria:

* Patients Requiring more than 3L/min of oxygen
* WHO progression scale = 5 to 8

Exclusion Criteria:

* Patients in 9 WHO progression class
* Patients with exclusion criteria to the CORIMUNO-19 cohort.
* Hypersensitivity to Bevacizumab or to any of their excipients.
* Pregnancy
* Active Cancer with undergoing treatment
* Oxygen patient requiring long-term oxygen before hospitalization
* Patient already included in a therapeutic trial; however, inclusion should be discussed case by case with the trial coordinator.
* Contraindication to bevacizumab, risk of bleeding especially hemoptysis, active venous or arterial thromboembolic disease and recent surgery.
* Hypersensitivity to the active substance or one of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of surviving patients without need for intubation for respiratory support | day 14

SECONDARY OUTCOMES:
Saturation of Oxygen in the blood (SaO2) | day 14
  value of a healthy individual occurs between 95 - 100
Arterial oxygen partial pressure (paO2) | day 14
  value of a healthy individual occurs between 75-100 mmHg
Ratio of arterial oxygen partial pressure to fractional inspired oxygen (paO2/FiO2) | day 14
  Normal level should be >500 Index of severity of acute respiratory distress syndrome (ARDS) mild if 200-300 moderate if 100-200 severe if < 200
CT-scan score | day 14
  based on a Likert scale with scores ranging from 1 to 5 (1-definitely no; 2-probably no; 3-equivocal; 4-probably yes; 5-definitely yes)
dyspnea | day 28
  measured on an visual analog scale (VAS), ranging from 0 (no dyspnea) to 10 (major dyspnea)
overall survival | day 14 and 28
admissionn to the intensive care unit (ICU) | day 14 and day 28
incidence of mechanical ventilation | day 14 and day 28
hospital length of stay | day 28
incidence of adverse event | day 28
VEGF plasma concentration | day 28

IPD SHARING:
Plan to Share IPD: Undecided